CLINICAL TRIAL: NCT00785161
Title: Penumbra Imaging Collaborative Study (PICS): A Multicenter Trial to Assess Outcome of Patients Revascularized by the Penumbra™ System
Brief Title: Penumbra Imaging Collaborative Study (PICS)
Acronym: PICS
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 1953.A
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Stroke
Keywords: Penumbra System; Mechanical Thrombectomy; Ischemic Stroke; Intervention; Neurovascular; Thrombus; Imaging; Ischemic Penumbra; Functional Outcome
MeSH Terms: conditions — Stroke; Ischemic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Penumbra System — Mechanical Thrombectomy in acute stroke

SUMMARY:
The primary aim of this study are to gather data on the "real world" experience of the Penumbra System and to determine if there is a correlate between the imaging-defined size of the ischemic penumbra at admission and patient outcome in patients already treated by the System. This will be accomplished by the collection of all available admission imaging data along with patient clinical and functional outcome results at 90-day follow-up to determine if a positive association exists between these variables. A secondary aim is to collect and summarize the 90-day functional outcome data for the purpose of sample size estimation for a potential randomized concurrent controlled trial. This will be accomplished by collecting the data on 90-day modified Rankin Scores (mRS) and all cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients who signed informed consent and revascularized by the Penumbra™ System in accordance to the Instruction For Use are eligible for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A stroke cohort who were revacularized by the Penumbra System
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an imaging-defined ischemic penumbra at admission that warrants revascularization by the Penumbra System. | Admission
Proportion of patients with successful revascularization of the occluded target vessel as defined by a TIMI score of 2 or 3 following use of the Penumbra System. | Post-Procedure
The proportion of patients with a modified Rankin Score (mRS) of ≤2 at 90 days post-procedure. | 90-Days Post-Procedure

SECONDARY OUTCOMES:
Neurological status as defined by the National Institute of Health Stroke Scale (NIHSS) scores at Admission and Discharge. | Admission and Discharge
Incidence of intracranial hemorrhage. | 24-Hours Post-Procedure
Incidence of device-related serious adverse events. | During the Procedure
All cause mortality at 90 days post-procedure. | 90-Days Post-Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Siu Po Sit, PhD, Study Director — Penumbra Inc.
Locations (1):
- Swedish Medical Center, Englewood, Colorado, United States

REFERENCES:
- See also: Penumbra Website — http://www.penumbrainc.com